CLINICAL TRIAL: NCT02048501
Title: Gut Hormone, Energy Expenditure and Body Composition Change in Subjects Who Succeed or Fail to Sustain Weight Loss After Roux-en-Y Gastric Bypass
Brief Title: Changes in Gut Hormones, Body Composition and Energy Expenditure After Roux-en-Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00049254
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Weight Loss
Keywords: Weight regain; Sustain weight loss; Weight loss; Gut hormones
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Basal Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Regain (Other): The weight regain group will include 20 subjects who underwent Roux-en-Y gastric bypass (RYGB) with a follow up of at least 2 years and have experienced excess weight loss (EWL) of at least 50% at 12 (+ 2) months post-operatively and regained at least 15% of the post-operative nadir weight.
  Interventions: Other: Resting Metabolic Rate (RMR); Other: Duel-energy x-ray absorptiometry (DEXA); Other: Visual Analog Scale (VAS); Other: Meal Stimulation Test
- Sustained Weight Loss (SWL) (Other): The sustained weight loss group will include 20 subjects who underwent Roux-en-Y gastric bypass (RYGB) with a follow up of at least 2 years and have experienced excess weight loss (EWL) of at least 50% at 12 (+ 2) months post-operatively and have regained less than 15% of the post-operative nadir weight.
  Interventions: Other: Resting Metabolic Rate (RMR); Other: Duel-energy x-ray absorptiometry (DEXA); Other: Visual Analog Scale (VAS); Other: Meal Stimulation Test

INTERVENTIONS:
Other: Resting Metabolic Rate (RMR) — Each subject will have their resting metabolic rate (RMR) measured. The RMR is assessed by indirect calorimetry measured with the metabolic cart. Oxygen consumption is converted into kilocalories. Subjects will be advised to avoid strenuous exercise for at least 48 hours prior to participation in the study and to sleep at least 6-8 hours the night before. Smoking and consuming caffeine will be prohibited 12 hours before the study begins.
Other: Duel-energy x-ray absorptiometry (DEXA) — During a separate appointment on the same day, or within 7 business days if same day is not possible, a body compositions analysis, including fat mass and fat free mass, will be assessed by dual-energy x-ray absorptiometry (DEXA), using a Hologic system.
  Other Names: Hologic Discovery A serial # 82364A version 13.3
Other: Visual Analog Scale (VAS) — Subjects will be asked to complete a 100-mm Visual Analog scale (VAS) to assess their appetite. The VAS will be completed prior to the meal stimulation test and at 30-minutes, 1-hour, 90 minutes and 2-hours after the meal. The VAS will contain questions assessing food intake, appetite, and hunger.
Other: Meal Stimulation Test — Subjects will consume a mixed-nutrient liquid meal 240-ml in 20 minutes. Prior to the meal stimulation test, a baseline 10-ml blood sample will be collected. The, during the meal stimulation test, 10-ml venous blood sample will be collected at 30 minute intervals up to two hours, for a total of 5 samples including the baseline sample. The blood samples will be used to measure fasting blood glucose, adipokines, myokines, gut hormones, amino acids, bile acids, vitamin B and vitamin D analysis with the appropriate assay method.

SUMMARY:
The purpose of this study is to gain a better understanding of the mechanism of weight regain through gut hormone (substances in the gut that control various functions of the digestive organs) and energy expenditure (the amount of energy a person uses to complete bodily activities).

Our hypothesis is that gut hormone response might be different among subjects who are able to maintain weight loss and subjects with weight regain.

For this study, investigators will measure fasting and postprandial (happening after a meal) gut hormones, bile acid, amino acids, vitamin B, vitamin D, myokines and adipokine levels in obese individuals who are at least 2 years after a Roux-en-Y gastric bypass (RYGB). Investigators will also measure resting metabolic rate (RMR) (the amount of energy expended daily) and body composition (the proportion of fat, muscle, and bone of an individual's body). The subjects body composition will be analyzed, including fat mass and fat free mass, by a Dual-Energy X-ray Absorptiometry (DEXA). This study will provide more information regarding the effect of RYGB on gut hormones, adipokines, bile acids, amino acids, and energy expenditure and body compositions.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years of age
2. Ability and willingness to provide informed consent

Exclusion Criteria:

1. Surgical/anatomical failure such as pouch enlargement, anastomosis dilation, formation of a gastrogastric fistula,
2. Currently on medication that might affect weight gain including GLP-1 analog
3. Inability to provide informed written consent.
4. Any known history of abnormal thyroid function.
5. Females who are pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Difference in pre and post-prandial plasma Glucagon-like peptide-1 (GLP-1) | Prior to meal stimulation test, 30 minutes, 60 minutes, 90 minutes and 120 after the meal stimulation test.
  The primary endpoints are a difference in pre postprandial plasma GLP-1 and PYY in subjects who underwent RYGB who succeed or fail to lose and maintain EWL goal.
Difference in pre and post-prandial Peptide YY (PYY) | Priot to the meal stimulation test, 30 minutes,60 minutes, 90 minutes, and 120 minutes after the meal stimulation test.
  The primary endpoints are a difference in pre postprandial plasma GLP-1 and PYY in subjects who underwent RYGB who succeed or fail to lose and maintain EWL goal.

CONTACTS AND LOCATIONS:
Overall Officials: Chan Park, MD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Metabolic and Weight Loss Surgery, Durham, North Carolina, United States